CLINICAL TRIAL: NCT00417521
Title: Pilot Study of Manualized Family Therapy for Adolescents With Anorexia Nervosa
Brief Title: Open Trial of Family-Based Treatment for Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4975R
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2006-12

CONDITIONS: Anorexia Nervosa
Keywords: Adolescents; Anorexia; Eating disorder; Family therapy
MeSH Terms: conditions — Anorexia Nervosa; Anorexia; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Family therapy (Experimental)
  Interventions: Behavioral: Family-Based Treatment

INTERVENTIONS:
Behavioral: Family-Based Treatment

SUMMARY:
This trial seeks to investigate the feasibility and effectiveness of delivering a newly manualized family-based treatment for adolescents with anorexia nervosa

DETAILED DESCRIPTION:
This open trial seeks to investigate the feasibility and effectiveness of delivering a newly manualized family-based treatment for adolescents with anorexia nervosa at a site beyond the treatment's origin. Adolescents ages 12-17 with anorexia nervosa or subthreshold anorexia nervosa were treated with up to one year of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-17
* Diagnosis of full or subthreshold anorexia nervosa
* At least one parent or guardian willing to participate in treatment

Exclusion Criteria:

* Bipolar Disorder, Psychotic Disorder, Substance Dependence
* Mental Retardation
* Acute suicidal risk
* Acute or unstable, poorly controlled chronic medical illness
* Weight below 75% ideal body weight

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2004-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
weight | end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Jones, Principal Investigator — New York State Psychiatric Institute